CLINICAL TRIAL: NCT03334760
Title: Breastfeeding and Complementary Feeding in Relation to BMI and Overweight at Ages 7 and 11 Years - a Path Analysis Within the Danish National Birth Cohort
Brief Title: Breastfeeding and Complementary Feeding in Relation to BMI and Overweight
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Camilla Schmidt Morgen, Project coordinator and primary investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: UHBispebjergFrederiksberg
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Child Overweight
Keywords: Cohort study; Infant feeding; Overweight; Child BMI; Breastfeeding; Intake of protein
MeSH Terms: conditions — Overweight; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Danish National Birth Cohort — DNBC is a nationwide cohort study of pregnant women and their offspring. The women were enrolled early during pregnancy between 1996 and 2002. They provided information on exposures during and after pregnancy by means of four computer-assisted telephone interviews in gestational weeks 12 and 30 and post-partum when the child was 6 and 18 months old.

SUMMARY:
This study examines the associations between different types of infant feeding and BMI and overweight in childhood. The study is based on the Danish National Birth Cohort, established in 1996.

DETAILED DESCRIPTION:
The objective of the study is to examine whether duration of breastfeeding, timing of introduction of complementary food and protein intake at 18 months are associated with BMI and overweight at ages 7 and 11 years, independent of BMI during infancy.

Children participating in the Danish National Birth Cohort were followed-up at ages 7 and 11years. Information on infant feeding, protein intake at 18 months, Ponderal Index at birth, child BMI (5 months, 12 months, 7 and 11 years) and several parental factors was available.

Path analysis was used to assess the direct and indirect effects of infant feeding on BMI z-scores at ages 7 (n= 36,481) and 11y (n=22,047). Logistic regression analyses were used to examine associations with overweight.

ELIGIBILITY:
Inclusion Criteria:

* The women were invited at their first antenatal visit at the general practitioner.Women were included if they intended to carry the pregnancy to term, had a permanent address in Denmark, and spoke Danish well enough to participate in telephone interviews.

Exclusion Criteria:

* Women who were not pregnant.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The DNBC was established during the years 1996 to 2003. A total of 100,418 pregnancies among a total of 92,274 women were enrolled into the cohort from all over Denmark. The women were invited at their first antenatal visit at the general practitioner. It is estimated that approximately 30% of all pregnant women in Denmark participated in the DNBC and the response rate is estimated to be 60%.The women were interviewed by telephone twice during their pregnancy, in approximately gestational week 16 (interview 1) and 31 (interview 2), and twice after their pregnancy when the child was approximately 6 (interview 3) and 18 months old (interview 4). During the computer assisted telephone interviews, the women gave detailed information on their physical and mental health, life style, nutrition and medicine use, and in the post-partum interviews the women gave information on growth, health and nutrition of the children.
Sampling Method: Non-Probability Sample
Enrollment: 100418 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Child overweight | 2003-2014
  The parent reported the height and weight of the children at approximately 7 and 11 years of age.

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the data from the DNBC may be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data are available.
Access Criteria: Researchers can apply the DNBC steering committee for data access.
URL: http://www.ssi.dk/Forskning/Forskningsomraader/Epidemiologi/BSMB

REFERENCES:
- [Derived] Morgen CS, Angquist L, Baker JL, Andersen AN, Sorensen TIA, Michaelsen KF. Breastfeeding and complementary feeding in relation to body mass index and overweight at ages 7 and 11 y: a path analysis within the Danish National Birth Cohort. Am J Clin Nutr. 2018 Mar 1;107(3):313-322. doi: 10.1093/ajcn/nqx058. PMID 29566190